CLINICAL TRIAL: NCT06264310
Title: A Phase 2, Double-Blind, Placebo-Controlled, Dose Range Finding Study to Assess Safety, Tolerability, Efficacy and Pharmacokinetics of the Relaxin Agonist R2R01 Combined With Standard of Care Versus Standard of Care Alone in Outpatients With Worsening Heart Failure (WHF)
Brief Title: To Evaluate the Safety, Tolerability and Efficacy of R2R01 Combined With SOC as Compared to SOC Alone in Outpatients With Worsening Heart Failure (WHF)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: River 2 Renal Corp. (Industry)
Collaborators: International HealthCare, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R2R01-WHF-201
Record Dates: First submitted 2024-01-31; First posted 2024-02-16 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-08

CONDITIONS: Heart Failure; Worsening Heart Failure (WHF)
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to one of four cohorts. Three groups will receive R2R01, and one group will receive placebo.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Treatment of all cohorts will be double-blind (all patients, study staff, investigators and Sponsor). Site pharmacist is unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): 8 study subjects will receive placebo once daily subcutaneous injection for 7 days.
  Interventions: Drug: Placebo
- 5.0 mg R2R01 (Experimental): 8 study subjects will receive 5.0 mg R2R01 once daily subcutaneous injection for 7 days.
  Interventions: Drug: R2R01
- 7.5 mg R2R01 (Experimental): 8 study subjects will receive 7.5 mg R2R01 once daily subcutaneous injection for 7 days.
  Interventions: Drug: R2R01
- 10.0 mg R2R01 (Experimental): 8 study subjects will receive 10.0 mg R2R01 once daily subcutaneous injection for 7 days.
  Interventions: Drug: R2R01

INTERVENTIONS:
Drug: Placebo — Matching placebo SC injection
  Arms: Placebo
Drug: R2R01 — Pharmaceutical Form: sterile 2R vials containing 10 mg of R2R01 for SC injection.
  Arms: 10.0 mg R2R01; 5.0 mg R2R01; 7.5 mg R2R01

SUMMARY:
This Study Aims to Evaluate the Safety, Tolerability and Efficacy of R2R01 Combined With SOC as Compared to SOC Alone in Outpatients With Worsening Heart Failure (WHF)

DETAILED DESCRIPTION:
This is a Phase 2, Double-Blind, Placebo-Controlled, Dose Range Finding Study to Assess Safety, Tolerability, Efficacy and Pharmacokinetics of the Relaxin Agonist R2R01 combined with Standard of Care versus Standard of Care Alone in Outpatients with Worsening Heart Failure (WHF). Each patient will undergo a screening period of up to 21 days, an active treatment period of 7 days, and a follow up period of 23 days after the last dose (30 days after the first dose), i.e., a total of up to 51 days total study duration.

This study is a four-parallel-cohort study. All patients will be randomized to one of the following Cohorts:

1. Cohort 1 (N=8): Placebo once daily SC for 7 days.
2. Cohort 2 (N=8): 5.0 mg R2R01 once daily SC for 7 days.
3. Cohort 3 (N=8): 7.5 mg R2R01 once daily SC for 7 days.
4. Cohort 4 (N=8): 10.0 mg R2R01 once daily SC for 7 days. All patients will present with worsening heart failure with congestion requiring SOC. The patient, in the opinion of the investigator, should be able to be treated for their symptoms without being admitted to the hospital. The planned 3-day hospitalization is to adequately manage any potential sign of hypotension and should not be required to treat the patient for the intensification of the diuretic therapy or same day IV loop diuretics. During the treatment period no new treatments for WHF should be initiated. This study will be conducted across approximately 8 centers in the US.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent, and able to follow instructions and comply with follow-up procedures.
2. History of symptomatic HF (heart failure).
3. Male or female ≥ 18 years of age at screening.
4. Previous hospitalization for HF within the last 12 months prior to screening.
5. Patients on optimal background therapy as per local practice for at least 30 days prior to screening and tolerating this well.
6. Patients must present with at least 2 of the following signs / symptoms of

   WHF congestion:
   1. Dyspnea
   2. Orthopnea
   3. Fatigue
   4. Jugular venous distension
   5. Rales
   6. Edema
7. Patient requires intensification (doubling the dose, adding another diuretic targeting another tubular segment) of oral diuretics, or IV diuresis for WHF as per Investigator at screening and treated as an outpatient patient.
8. Estimated Glomerular Filtration Rate (eGFR) between 20 and 75 mL/ min/1.73 m2 (calculated using the CKD-EPI equation) at screening.
9. NT-pro-BNP levels at screening:

   1. ≥ 1000 pg/mL for patients with LVEF ≤ 40%
   2. ≥ 700 pg/mL for patients with LVEF > 40%
   3. ≥ 1500 pg/mL for patients with current atrial fibrillation, regardless of LVEF. For patients with BMI ≥ 30 kg/m2 the NT-pro-BNP values are lowered by 20%. The values are as follows:

   <!-- -->

   1. ≥ 800 pg/mL for patients with LVEF ≤ 40%
   2. ≥ 560 pg/mL for patients with LVEF > 40%
   3. ≥ 1200 pg/mL for patients with current atrial fibrillation, regardless of LVEF. The most recent LVEF value assessed in the 12 months prior to screening should be used.
10. Systolic Blood Pressure (SBP) ≥ 105 mmHg at screening.
11. Willing and able to stay in the clinic for observation/monitoring for 3 days.
12. Willing to self-administer all SC injections.

Exclusion Criteria:

1. Patients with blood pressure > 180 mmHg or persistent heart rate > 130 bpm at Screening.
2. History of symptomatic hypotension.
3. History of orthostatic hypotension.
4. Temperature > 38.5°C (oral or equivalent) or sepsis or active infection requiring antimicrobial treatment.
5. Clinical evidence of acute coronary syndrome (ACS) currently or within 30 days prior to Screening.
6. Acute Heart Failure (AHF) due to significant arrhythmias, which include any of the following: sustained ventricular tachycardia, bradycardia with sustained ventricular rate < 45 bpm or atrial fibrillation/flutter with sustained ventricular response of > 130 bpm.
7. The daily use of IV or oral steroids (including but not limited to the use of IV or oral steroids for respiratory disorders or COPD). Note, inhaled steroids are allowed.
8. IV antimicrobial treatment for sepsis or active infection.
9. Patients with severe renal impairment defined at Screening eGFR < 20 mL/min/1.73m2 (calculated using the CKD-EPI Equation), and/or those receiving current or planned dialysis or ultrafiltration.
10. Patients with hemoglobin < 10 g/dL, or a history of blood transfusion within the 14 days prior to screening, or active life-threatening gastrointestinal bleeding.
11. Known hepatic impairment (as evidenced by total bilirubin > 3 mg/dL, or increased ammonia levels, if performed) or history of cirrhosis with evidence of portal hypertension such as varices.
12. Significant, uncorrected, left ventricular outflow obstruction, such as obstructive hypertrophic cardiomyopathy or severe aortic stenosis (i.e., aortic valve area < 1.0 cm2 or mean gradient > 40 mmHg on echocardiogram), and/or severe mitral stenosis.
13. Severe aortic insufficiency or severe mitral regurgitation for which surgical or percutaneous intervention is indicated.
14. Documented, prior to or at the time of screening, restrictive amyloid myocardiopathy, or acute myocarditis or hypertrophic obstructive, restrictive, or constrictive cardiomyopathy.
15. Any major solid organ transplant recipient or planned/ anticipated organ transplant within 1 year.
16. Major surgery, including implantable devices (e.g., implantable cardioverter defibrillator, cardiac resynchronization therapy), or major neurologic event including cerebrovascular events, within 30 days prior to screening.
17. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past year with a current life expectancy less than 1 year due to the malignancy.
18. Pregnant or nursing (lactating) women, where pregnancy was defined as the state of a female after conception and until the termination of gestate, confirmed by a positive human chorionic gonadotropin laboratory test.
19. Use of other investigational drugs within 30 days prior to Screening.
20. History of known hypersensitivity/prior exposure to R2R01 or serelaxin.
21. Any other medical condition(s) that might put the patient at risk or influence study results in the Investigator's opinion, or that the Investigator deems unsuitable for the study including drug or alcohol abuse or psychiatric, behavioral, or cognitive disorders sufficient to interfere with the patient's ability to understand and comply with the protocol instructions or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-11-04 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Number and rate of patients with one or more TEAEs (treatment emergent AE's) and/or serious TEAEs as assessed by CTCAE v5.0. | Day 7, Day 30
  To assess the safety and tolerability of various dose levels of R2R01 in WHF patients at Day 7 and Day 30.
Number and rate of patients with one or more TEAEs (treatment emergent AE's) and/or serious TEAEs as assessed by CTCAE v5.0. | Day 30
  To select the appropriate dose for Study R2R01-WHF-202

SECONDARY OUTCOMES:
Change from Baseline on NT-pro-BNP using descriptive and summary statistics by dose level at Day 7 and Day 30. | Day 7, Day 30
  To evaluate the effect of R2R01 on NT-pro-BNP as a proxy for cardiac congestion at Day 7 and Day 30.
Change from baseline on Cystatin C and creatinine clearance using descriptive and summary statistics by dose level at Day 7 and Day 30. | Day 7, Day 30
  To evaluate the effect of R2R01 on Cystatin C and creatinine clearance (eGFR using CKD-EPI Equation using both creatinine and cystatin C) at Day 7 and Day 30.
Number of patients requiring dose adjustment of oral diuretics during the 30-day follow-up. | Day 30
  To evaluate the effect of R2R01 on therapy with diuretics at Day 30.
Number of patients with an event of: WHF-induced SDAC or other outpatient clinic visits requiring additional intensification of the therapy/IV loop diuretics using descriptive and summary statistics for change from baseline by dose level at Day 30. | Day 30
  To evaluate the effect of R2R01 at Day 30 on:
  WHF-induced Same Day Access Clinic (SDAC)--or other outpatient clinic visits requiring, additional intensification of the therapy/IV loop diuretics.
Number of cardiovascular hospitalizations among patients using descriptive and summary statistics for change from baseline by dose level at Day 30. | Day 30
  To evaluate the effect of R2R01 at Day 30 on: Cardiovascular (CV) hospitalizations.
Number of all-cause hospitalizations among patients using descriptive and summary statistics for change from baseline by dose level at Day 30. | Day 30
  To evaluate the effect of R2R01 at Day 30 on: All-cause hospitalizations.
Number of patients with CV mortality using descriptive and summary statistics for change from baseline by dose level at Day 30. | Day 30
  To evaluate the effect of R2R01 at Day 30 on: CV mortality.
Number of patients with all-cause mortality using descriptive and summary statistics for change from baseline by dose level at Day 30. | Day 30
  To evaluate the effect of R2R01 at Day 30 on: All-cause mortality.

CONTACTS AND LOCATIONS:
Locations (18):
- United States (14):
  - Mayo Clinic, Phoenix, Arizona
  - California Pacific Medical Center, San Francisco, California
  - Mayo Clinic, Jacksonville, Florida
  - Piedmont Hospital Transplant, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - VA North Texas Health Care, Dallas, Texas
  - Baylor Scott and White All Saints Medical Center, Fort Worth, Texas
- Germany (2):
  - University of Duisburg-Essen, Essen, North Rhine-Westphalia
  - University of Munster, Münster, North Rhine-Westphalia
- Italy (2):
  - University of Bologna, Bologna
  - University-Hospital of Padova, Padua

IPD SHARING:
Plan to Share IPD: No